CLINICAL TRIAL: NCT04082026
Title: Towards an Evidence-based Scalable Psychological Intervention for Young Adolescents: Feasibility cRCT of Group Psychological Help for Young Burundian Refugee Adolescents in Tanzania.
Brief Title: Early Adolescent Skills for Emotions Tanzania Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Rescue Committee (Other)
Collaborators: World Health Organization (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYPD 1.00.003
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: The research study compared the EASE treatment (7 weekly sessions for adolescents and 3 for their caregivers) against an Enhanced Treatment as Usual (ETAU) consisting of a single psychoeducation individual session, jointly for eligible adolescents and their caregivers. ETAU included information on: (i) the results of the screening; (ii) self-care strategies; and, (iii) seeking services from local health or community services offering psychosocial / mental health care support.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Adolescent Skills for Emotions (EASE) (Experimental): EASE has four core features: Seven group sessions for young adolescents and three for their caregivers; Delivered by non-specialists; Trans-diagnostic: addressing depression, anxiety, distress, and other problems as defined by the young people themselves; and Designed for young people and their caregivers in low- and middle-income countries living in communities affected by adversity.
  Interventions: Behavioral: Early Adolescent Skills for Emotions EASE)
- Enhanced Treatment As Usual (ETAU) (Placebo Comparator): The Enhanced Treatment as Usual (ETAU) consisted of a single psychoeducation individual session, jointly for eligible adolescents and their caregivers, that included information on: (i) the results of the screening; (ii) self-care strategies; and, (iii) seeking services from local health or community services offering psychosocial / mental health care support.
  Interventions: Behavioral: Early Adolescent Skills for Emotions EASE)

INTERVENTIONS:
Behavioral: Early Adolescent Skills for Emotions EASE) — EASE is conducted in 7 weekly group sessions with adolescents. EASE sessions help adolescents:
  * Identify their feelings and body reactions
  * Practice breathing exercises
  * Get active: Make a plan to positively change their actions
  * Manage their problems
  Other Names: Enhanced Treatment as Usual (ETAU)

SUMMARY:
The goal of this pilot is to test the World Health Organization (WHO) Early Adolescent Skills for Emotions intervention, a new psychological intervention. The pilot in Tanzania adapted the manual for young adolescent Burundian refugees in Tanzania (ages 10 - 14) with prolonged disabling distress living in communities affected by adversity. We conducted a formative study to adapt the EASE material, followed by small feasibility RCT (M=72) along with a process evaluation.

DETAILED DESCRIPTION:
WHO is developing a set of scalable brief psychological programs: a new generation of shorter, less expensive and trans-diagnostic programs that can be delivered by non-specialized providers (e.g. without formal education or experience in mental health), to reduce common mental health symptoms and improve psychosocial functioning. In this pilot in Tanzania, the IRC, JHU and WHO seek to assess EASE, a much needed, brief psychological intervention developed specifically for young adolescents and their caregivers, and applicable in different humanitarian contexts.

The IRC, JHU and WHO, in collaboration with UNHCR, Muhimbili University of Health and Allied Sciences in Tanzania, and Village Health Works , adapted and contextualized the EASE intervention for Burundian refugee young adolescents in Tanzania. The adaptation had three steps:

First, the IRC conducted a desk review focusing on the cultural context for mental health research among Burundian refugees, covering local concepts, beliefs and practices associated with psychosocial support.

Second, the IRC conducted a formative qualitative study, consisting of 88 semi-structured qualitative interviews (free listing (n=61) and key informant interviews (n=25)), including with Burundian adolescent boys and girls (See Tables 1 & 2 in Annex for breakdown of interview participants). This was followed by four focus group discussions (n=20) using cognitive interviewing techniques with adolescents and caregivers to seek feedback specifically on example intervention materials.

Third, the IRC and its partners used findings from the desk review and the qualitative study to inform an adaptation workshop in May 2018 held in Kibondo, Tanzania. For the adaptation workshop, the IRC convened the WHO, IRC mental health field staff, Village Health Works staff, and Dr Samuel Likindikoki from the Muhimbili University of Health and Allied Sciences. The adaptation workshop included a review of the data collected during the ethnographic study, as well as a mock run-through of the EASE materials, which allowed for an in-depth review of the intervention content.

The EASE pilot implementation and testing phase had eight main activities: 1) initial screening of adolescents for eligibility into the EASE program; 2) baseline data collection with the eligible participants and caregivers; 3) facilitator training; 4) development of a referral protocol to ensure adequate services for participants who experienced violence or were at high risk of suicide; 5) implementation of the EASE sessions; 6) implementation of the "Enhanced treatment as usual" sessions (our control condition, conducted at the same time as the EASE sessions); 7) endline data collection; and 8) process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* a score of eight or more points on the Child Psychosocial Distress Screener (CPDS)

Exclusion Criteria:

* High suicide risk
* Severe impairment
* Lack of parental consent

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
African Youth Psychosocial Assessment | 2 months
  Adolescent psychological distress was assessed using the total problem score from the African Youth Psychosocial Assessment (AYPA), which consists of 33 items capturing internalizing symptoms, externalizing symptoms, and somatic complaints with a 4-point response scale (range 0-99). The AYPA also includes a subscale capturing prosocial behaviors (8 items, range 0-24). While we relied on the adolescent-reported AYPA as our primary outcome, we also included a caregiver-reported version of the AYPA to allow for comparison.

SECONDARY OUTCOMES:
Short Warwick-Edinburgh Mental Wellbeing Scale | 2 months
  Adolescent mental well-being was assessed with the 14-item Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS; 5-point response scale, range 0-28) (Tennant et al., 2007).
Child Post Traumatic Stress Disorder (PTSD) Symptom Scale | 2 months
  Adolescent PTSD symptoms were assessed with the Child PTSD Symptom Scale (CPSS) (Foa, Johnson, Feeny, & Treadwell, 2001). This 17-item measure uses a 4-point response scale to assess PTSD symptoms according to Diagnostic and Statistical Manual of Mental Disorders criteria (range 0-51).
Child Trauma Questionnaire (CTQ) | 2 months
  Adolescent traumatic exposures were measured using a 15-item version of the Child Trauma Questionnaire (CTQ) that was adapted locally (5-point response scale, range 0-60) (Bernstein & Fink, 1998; Charak, de Jong, Berckmoes, Ndayisaba, & Reis, 2017).
Adolescent Exposure to Violence | 2 months
  Adolescent exposure to violence was examined using a locally developed list of 33 dichotomous items (yes or no) that assessed lifetime experiences of violence perpetrated both by caregivers and non-caregivers (including emotional, physical, and sexual abuse). Follow-up questions to each item determined recency of violence (i.e., whether or not it had occurred within the past two months).

CONTACTS AND LOCATIONS:
Locations (1):
- International Rescue Committee, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No